CLINICAL TRIAL: NCT04174547
Title: An Integrated European Platform to Conduct Translational Studies in Myelodysplastic Syndromes Based on the EuroBloodNet Infrastructure
Brief Title: An European Platform for Translational Research in Myelodysplastic Syndromes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: TRS-2018-00000745
Record Dates: First submitted 2019-11-12; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Myelodysplastic Syndromes
Keywords: Somatic mutations; Clonal hematopoiesis; Biomarkers; Immune escape; Innovative predictive models; EuroBloodNet
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Peripheral blood and marrow samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Clonal hematopoiesis (AIM 1): The investigators will analyze the genomic features of clonal dominance and ineffective hematopoiesis in elderly subjects enrolled in two population-based studies: "Health and Anemia" study [Haematologica 2010;95:1849], and "Monzino 80-plus" study [BMC Neurol.2011;11:54, validation cohort]. Overall in 5000 subjects aged >65y peripheral blood samples (in some cases collected at different time points) will be available for biological investigations.
- Innovative predictive models in MDS (AIM2): The investigators will base on large retrospectove adult MDS population with comprehensive genomic and clinical data available within EuroBloodNet network (data on 3000 patients will be available), to accurately predict clinical outcomes in MDS at individual-patient level.
  The investigators plan to define 2 homogenous clinical cohorts (learning and testing cohort at 2:1 ratio) in order to define distinct patterns and genetic groups within MDS and to independently validate their predictive value.
- Predictive biomarkers in MDS (AIM3): The investigators will analyze MDS patients enrolled in prospective clinical trials conducted within the EuroBloodNet network. Overall 350 patients treated with azacitidine from prospective studies (VidazaAllotrial, RELAZA02 trial, AZA-Ida study, intensive AZA study) will be available for biological investigations to define biomarkers associated with clinical response. Validation of biomarkers will then be performed in an independent cohort including 320 patients (AZA-PLUS trial). In all these studies, biobanking of bone marrow (BM) and peripheral blood (PB) samples has been systematically performed, providing a unique resource to be investigated within this proposal.

SUMMARY:
Rationale Myelodysplastic syndromes (MDS) are rare cancers with unmet medical needs. Study of MDS has been rapidly transformed by genome characterization.

The investigators hypothesize that comprehensive analyses of large patient population will allow to correctly estimate the effect of each mutation on clinical outcomes, and that niche factors and immune dysfunctions may influence the development of MDS, clonal evolution and response to treatments

Aims

1- Investigate gene mutations, niche factors and immune dysfunctions influencing the development of MDS, and define biomarkers for early identification of individuals at risk; 2- Develop prognostic models for MDS patients through integration of comprehensive genomic/clinical information; 3- Define biomarkers to better stratify the individual probability of response to specific treatments

Methods EuroBloodNet, the European Reference Network in rare hematological diseases, will provide a basis for research activities. Study of genomic features of clonal dominance in elderly subjects enrolled in large population-based studies and description of the dynamics of clonal establishment and evolution; study of bone marrow microenvironment to identify immune dysfunctions influencing MDS development. Development of inclusive statistical models to accurately predict clinical outcome at individual level, based on large MDS populations with comprehensive genomic/clinical data. Finally, analysis of mutational screening and immune profiles from patients enrolled in prospective trials, to provide evidence on genetic/immunologic profiles associated with probability of response to specific compounds

Expected results To characterize how clonal hematopoiesis relates to the induction of MDS clinical phenotype, and to test the utility of gene sequencing to detect subjects at risk of developing MDS. To define effective prognostic systems and biomarkers to stratify the individual probability of response to treatment

DETAILED DESCRIPTION:
MDS typically occurs in elderly people and a portion of these subjects evolve into acute myeloid leukemia (AML). The natural history of MDS is highly heterogeneous, and therefore a risk-adapted treatment strategy is mandatory.

The presence of mutations in a given individual has only limited predictive power, as conversion to MDS is rare regardless of mutation status. In addition, in patients with overt MDS, genetic abnormalities explain only a proportion of the total hazard for survival, meaning that a large percentage is still associated with clinical and non-mutational factors. Comprehensive analyses of large patient populations are warranted to correctly estimate the independent effect of each mutation on clinical outcome and response to treatment.

Moreover, environmental factors influencing the development of MDS and the probability of response to specific treatments are to be characterized. They include alterations in the immune system. In this context, a significant association was found between autoimmune disorders and MDS, and activation of the inflammasome may contribute to MDS development

AIMS 1- Investigate gene mutations, niche factors and immune dysfunctions influencing the development of MDS, and define biomarkers for early identification of individuals at risk; 2- Develop prognostic models for MDS patients through integration of comprehensive genomic/clinical information; 3- Define biomarkers to better stratify the individual probability of response to specific treatments

EXPERIMENTAL DESIGN

AIM1

1a) The investigators will analyze the genomic features of clonal dominance and ineffective hematopoiesis in elderly subjects enrolled in different population-based studies.

Peripheral blood samples will be available for biological investigations. A low-cost, high-throughput platform for mutation screening of 72 genes known to be relevant in MDS will be used.

1b) In order to gain further insight into the MDS genetic heterogeneity, the investigators will perform DNA sequencing in hematopoietic progenitors single cells to clarify the clonal architecture of marrow dysplasia in HSC, the dynamics of clonal establishment and expansion during hematopoietic differentiation, and their relationship with the disease phenotype and evolution

1c) In selected elderly individuals, the investigators will study the transcriptome (RNA sequencing) of isolated mesenchymal stromal cells (MSC) and marrow microenvironment (i.e., innate ad adaptive immunity) with the aim to identify niche factors that may influence the development of a MDS phenotype in elderly subjects with clonal hematopoiesis. Moreover, in patients suffering from both MDS and autoimmune disorder, the investigators will analyze immunological parameters. They will be compared with those of patients with MDS but without immune disorder, and patients with immune disorders without MDS

AIM2

In myeloid malignancies, it was shown that large knowledge banks of matched genomic-clinical data can improve clinical decision-making.

In the present project, basing on large MDS populations with comprehensive genomic and clinical data available within EuroBloodNet network (data on >3000 patients will be available), the investigators will develop inclusive, multistage statistical models (Bayesian network analysis and clustering) to accurately predict clinical outcomes in MDS at individual-patient level. The investigators plan to define 2 homogenous clinical cohorts in order to define distinct patterns and genetic groups within MDS and to independently validate their predictive value. As a research tool, the investigators plan to create a prototype portal within our EuroBloodNet website that allows outcome predictions to be generated based on this data set for user-defined constellations of genomic features and clinical variables. The reliability of this tool on clinical decision making will be tested in a prospective observational trial in the context of EuroBloodNet

AIM3

The investigators will analyze the mutational status and immune landscape associated with response to HMA in MDS patients enrolled in prospective clinical trials conducted within the EuroBloodNet network. Patients treated with azacitidine from prospective studies will be available for biological investigations to define biomarkers associated with clinical response. Validation of biomarkers will then be performed in an independent cohort. In all these studies, biobanking of bone marrow (BM) and peripheral blood (PB) samples has been systematically performed, providing a unique resource to be investigated within this proposal. Data on mutational screening and immune profiles are already available in most patients, and were obtained by comparable methods. For mutation screening, a NGS approach covering key genes involved in myeloid malignancies and the response to HMA was used. For a comprehensive immunological characterization of T lymphocytes, NK cells and ILC cells, standardized flow cytometric protocols were used, which will provide novel insights into frequency, differentiation and activity of these cells in response to therapy. Complementary immunoassays based on Luminex technology will be used to quantify secretory proteins (cytokines, chemokines, growth factors) in BM and PB plasma samples.

ELIGIBILITY:
AIM 1

Inclusion Criteria:

- Individuals aged 65 years or older from population-based studies (retrospective cohort)

Exclusion Criteria:

- lack of biological samples availability

AIM 2

Inclusion Criteria:

- adults patients (>18 years) with a diagnosis of MDS according to WHO criteria (retrospective cohort)

Exclusion Criteria:

- lack of availability of information on clinical and DNA mutational screening data

AIM 3

Inclusion Criteria:

- adults patients (>18 years) with a diagnosis of MDS according to WHO criteria and treated with HMAs

Exclusion Criteria:

- lack of biological samples availability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AIM 1 Individuals enrolled in the population-based "Health and Anemia" and "Monzino 80+" studies, with biological samples available at prevalence day
  AIM 2 Patients receiving a diagnosis of MDS within EuroBloodNet clinical network, for which complete information on clinical and DNA mutational screening data is available
  AIM 3
  * Testing cohort: MDS patients treated with HMAs within prospective clinical trials (VidazaAllotrial, RELAZA02 trial, AZA-Ida study, intensive AZA study), with biological samples availability
  * Validation cohort: adults MDS patients treated with HMAs within the prospective clinical trial AZA-PLUS, with biological samples availability
Sampling Method: Non-Probability Sample
Enrollment: 8670 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
DNA mutations in hematopoietic cells | 0-24 months
  The investigotors will study the prevalence and type of somatic mutations by a low-cost, high-throughput platform including 72 genes, relevant in myeloid neoplasms.
RNA expression on hematopoietic progenitors and mesenchymal stromal cells | 6-24 months
  The investigators will study the genes diffentially expressed between cell populations of interest and normal controls
Predictive biomarkers for survival and response to treatment | 0-30 months
  The investigators will define, by innovative bayesian and clustering models, independent clinical and molecular factors associated to the probability of survival and response to specific treatments.
Frequency and function of T lymphocytes, NK cells and ILC cells | 6-30 motnhs
  The investigators will analyse by flow-cytometry the frequency of T lymphocytes, NK cells and ILC cells during different disease stages and in response to therapy.
  Complementary immunoassays based on Luminex technology will be used to quantify secretory proteins (cytokines, chemokines, growth factors).

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Della Porta, MD, Principal Investigator — HUMANITAS Cancer Center
Locations (4):
- Service d'hématologie séniors - Hôpital St Louis / Université Paris 7, Paris, France
- University of Leipzig Medical Center, Leipzig, Germany
- Istituto Clinico Humanitas, Rozzano, Milan, Italy
- Josep Carreras Leukaemia Research Institute (IJC), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ades L, Itzykson R, Fenaux P. Myelodysplastic syndromes. Lancet. 2014 Jun 28;383(9936):2239-52. doi: 10.1016/S0140-6736(13)61901-7. Epub 2014 Mar 21. PMID 24656536
- [Background] Malcovati L, Hellstrom-Lindberg E, Bowen D, Ades L, Cermak J, Del Canizo C, Della Porta MG, Fenaux P, Gattermann N, Germing U, Jansen JH, Mittelman M, Mufti G, Platzbecker U, Sanz GF, Selleslag D, Skov-Holm M, Stauder R, Symeonidis A, van de Loosdrecht AA, de Witte T, Cazzola M; European Leukemia Net. Diagnosis and treatment of primary myelodysplastic syndromes in adults: recommendations from the European LeukemiaNet. Blood. 2013 Oct 24;122(17):2943-64. doi: 10.1182/blood-2013-03-492884. Epub 2013 Aug 26. PMID 23980065
- [Background] Greenberg PL, Tuechler H, Schanz J, Sanz G, Garcia-Manero G, Sole F, Bennett JM, Bowen D, Fenaux P, Dreyfus F, Kantarjian H, Kuendgen A, Levis A, Malcovati L, Cazzola M, Cermak J, Fonatsch C, Le Beau MM, Slovak ML, Krieger O, Luebbert M, Maciejewski J, Magalhaes SM, Miyazaki Y, Pfeilstocker M, Sekeres M, Sperr WR, Stauder R, Tauro S, Valent P, Vallespi T, van de Loosdrecht AA, Germing U, Haase D. Revised international prognostic scoring system for myelodysplastic syndromes. Blood. 2012 Sep 20;120(12):2454-65. doi: 10.1182/blood-2012-03-420489. Epub 2012 Jun 27. PMID 22740453
- [Background] Schanz J, Tuchler H, Sole F, Mallo M, Luno E, Cervera J, Granada I, Hildebrandt B, Slovak ML, Ohyashiki K, Steidl C, Fonatsch C, Pfeilstocker M, Nosslinger T, Valent P, Giagounidis A, Aul C, Lubbert M, Stauder R, Krieger O, Garcia-Manero G, Faderl S, Pierce S, Le Beau MM, Bennett JM, Greenberg P, Germing U, Haase D. New comprehensive cytogenetic scoring system for primary myelodysplastic syndromes (MDS) and oligoblastic acute myeloid leukemia after MDS derived from an international database merge. J Clin Oncol. 2012 Mar 10;30(8):820-9. doi: 10.1200/JCO.2011.35.6394. Epub 2012 Feb 13. PMID 22331955
- [Background] Nomdedeu M, Calvo X, Pereira A, Carrio A, Sole F, Luno E, Cervera J, Vallespi T, Munoz C, Gomez C, Arias A, Such E, Sanz G, Grau J, Insunza A, Calasanz MJ, Ardanaz MT, Hernandez-Rivas JM, Azaceta G, Alvarez S, Sanchez J, Martin ML, Bargay J, Gomez V, Cervero CJ, Allegue MJ, Collado R, Campo E, Esteve J, Nomdedeu B, Costa D; Spanish Group of Myelodysplastic Syndromes. Prognostic impact of chromosomal translocations in myelodysplastic syndromes and chronic myelomonocytic leukemia patients. A study by the spanish group of myelodysplastic syndromes. Genes Chromosomes Cancer. 2016 Apr;55(4):322-7. doi: 10.1002/gcc.22333. Epub 2015 Dec 22. PMID 26690722
- [Background] Schanz J, Tuchler H, Sole F, Mallo M, Luno E, Cervera J, Grau J, Hildebrandt B, Slovak ML, Ohyashiki K, Steidl C, Fonatsch C, Pfeilstocker M, Nosslinger T, Valent P, Giagounidis A, Aul C, Lubbert M, Stauder R, Krieger O, Le Beau MM, Bennett JM, Greenberg P, Germing U, Haase D. Monosomal karyotype in MDS: explaining the poor prognosis? Leukemia. 2013 Oct;27(10):1988-95. doi: 10.1038/leu.2013.187. Epub 2013 Jun 21. PMID 23787396
- [Background] Valcarcel D, Adema V, Sole F, Ortega M, Nomdedeu B, Sanz G, Luno E, Canizo C, de la Serna J, Ardanaz M, Marco V, Collado R, Grau J, Montoro J, Mallo M, Vallespi T. Complex, not monosomal, karyotype is the cytogenetic marker of poorest prognosis in patients with primary myelodysplastic syndrome. J Clin Oncol. 2013 Mar 1;31(7):916-22. doi: 10.1200/JCO.2012.41.6073. Epub 2013 Jan 14. PMID 23319689
- [Background] Della Porta MG, Alessandrino EP, Bacigalupo A, van Lint MT, Malcovati L, Pascutto C, Falda M, Bernardi M, Onida F, Guidi S, Iori AP, Cerretti R, Marenco P, Pioltelli P, Angelucci E, Oneto R, Ripamonti F, Bernasconi P, Bosi A, Cazzola M, Rambaldi A; Gruppo Italiano Trapianto di Midollo Osseo. Predictive factors for the outcome of allogeneic transplantation in patients with MDS stratified according to the revised IPSS-R. Blood. 2014 Apr 10;123(15):2333-42. doi: 10.1182/blood-2013-12-542720. Epub 2014 Feb 20. PMID 24558201
- [Background] Papaemmanuil E, Gerstung M, Malcovati L, Tauro S, Gundem G, Van Loo P, Yoon CJ, Ellis P, Wedge DC, Pellagatti A, Shlien A, Groves MJ, Forbes SA, Raine K, Hinton J, Mudie LJ, McLaren S, Hardy C, Latimer C, Della Porta MG, O'Meara S, Ambaglio I, Galli A, Butler AP, Walldin G, Teague JW, Quek L, Sternberg A, Gambacorti-Passerini C, Cross NC, Green AR, Boultwood J, Vyas P, Hellstrom-Lindberg E, Bowen D, Cazzola M, Stratton MR, Campbell PJ; Chronic Myeloid Disorders Working Group of the International Cancer Genome Consortium. Clinical and biological implications of driver mutations in myelodysplastic syndromes. Blood. 2013 Nov 21;122(22):3616-27; quiz 3699. doi: 10.1182/blood-2013-08-518886. Epub 2013 Sep 12. PMID 24030381
- [Background] Papaemmanuil E, Cazzola M, Boultwood J, Malcovati L, Vyas P, Bowen D, Pellagatti A, Wainscoat JS, Hellstrom-Lindberg E, Gambacorti-Passerini C, Godfrey AL, Rapado I, Cvejic A, Rance R, McGee C, Ellis P, Mudie LJ, Stephens PJ, McLaren S, Massie CE, Tarpey PS, Varela I, Nik-Zainal S, Davies HR, Shlien A, Jones D, Raine K, Hinton J, Butler AP, Teague JW, Baxter EJ, Score J, Galli A, Della Porta MG, Travaglino E, Groves M, Tauro S, Munshi NC, Anderson KC, El-Naggar A, Fischer A, Mustonen V, Warren AJ, Cross NC, Green AR, Futreal PA, Stratton MR, Campbell PJ; Chronic Myeloid Disorders Working Group of the International Cancer Genome Consortium. Somatic SF3B1 mutation in myelodysplasia with ring sideroblasts. N Engl J Med. 2011 Oct 13;365(15):1384-95. doi: 10.1056/NEJMoa1103283. Epub 2011 Sep 26. PMID 21995386
- [Background] Della Porta MG, Tuechler H, Malcovati L, Schanz J, Sanz G, Garcia-Manero G, Sole F, Bennett JM, Bowen D, Fenaux P, Dreyfus F, Kantarjian H, Kuendgen A, Levis A, Cermak J, Fonatsch C, Le Beau MM, Slovak ML, Krieger O, Luebbert M, Maciejewski J, Magalhaes SM, Miyazaki Y, Pfeilstocker M, Sekeres MA, Sperr WR, Stauder R, Tauro S, Valent P, Vallespi T, van de Loosdrecht AA, Germing U, Haase D, Greenberg PL, Cazzola M. Validation of WHO classification-based Prognostic Scoring System (WPSS) for myelodysplastic syndromes and comparison with the revised International Prognostic Scoring System (IPSS-R). A study of the International Working Group for Prognosis in Myelodysplasia (IWG-PM). Leukemia. 2015 Jul;29(7):1502-13. doi: 10.1038/leu.2015.55. Epub 2015 Feb 27. PMID 25721895
- [Background] Della Porta MG, Travaglino E, Boveri E, Ponzoni M, Malcovati L, Papaemmanuil E, Rigolin GM, Pascutto C, Croci G, Gianelli U, Milani R, Ambaglio I, Elena C, Ubezio M, Da Via' MC, Bono E, Pietra D, Quaglia F, Bastia R, Ferretti V, Cuneo A, Morra E, Campbell PJ, Orazi A, Invernizzi R, Cazzola M; Rete Ematologica Lombarda (REL) Clinical Network. Minimal morphological criteria for defining bone marrow dysplasia: a basis for clinical implementation of WHO classification of myelodysplastic syndromes. Leukemia. 2015 Jan;29(1):66-75. doi: 10.1038/leu.2014.161. Epub 2014 May 20. PMID 24935723
- [Background] Della Porta MG, Jackson CH, Alessandrino EP, Rossi M, Bacigalupo A, van Lint MT, Bernardi M, Allione B, Bosi A, Guidi S, Santini V, Malcovati L, Ubezio M, Milanesi C, Todisco E, Voso MT, Musto P, Onida F, Iori AP, Cerretti R, Grillo G, Molteni A, Pioltelli P, Borin L, Angelucci E, Oldani E, Sica S, Pascutto C, Ferretti V, Santoro A, Bonifazi F, Cazzola M, Rambaldi A. Decision analysis of allogeneic hematopoietic stem cell transplantation for patients with myelodysplastic syndrome stratified according to the revised International Prognostic Scoring System. Leukemia. 2017 Nov;31(11):2449-2457. doi: 10.1038/leu.2017.88. Epub 2017 Mar 21. PMID 28321120
- [Background] Jaiswal S, Fontanillas P, Flannick J, Manning A, Grauman PV, Mar BG, Lindsley RC, Mermel CH, Burtt N, Chavez A, Higgins JM, Moltchanov V, Kuo FC, Kluk MJ, Henderson B, Kinnunen L, Koistinen HA, Ladenvall C, Getz G, Correa A, Banahan BF, Gabriel S, Kathiresan S, Stringham HM, McCarthy MI, Boehnke M, Tuomilehto J, Haiman C, Groop L, Atzmon G, Wilson JG, Neuberg D, Altshuler D, Ebert BL. Age-related clonal hematopoiesis associated with adverse outcomes. N Engl J Med. 2014 Dec 25;371(26):2488-98. doi: 10.1056/NEJMoa1408617. Epub 2014 Nov 26. PMID 25426837
- [Background] Weidner H, Rauner M, Trautmann F, Schmitt J, Balaian E, Mies A, Helas S, Baschant U, Khandanpour C, Bornhauser M, Hofbauer LC, Platzbecker U. Myelodysplastic syndromes and bone loss in mice and men. Leukemia. 2017 Apr;31(4):1003-1007. doi: 10.1038/leu.2017.7. Epub 2017 Jan 11. No abstract available. PMID 28074069
- [Background] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Finelli C, Giagounidis A, Schoch R, Gattermann N, Sanz G, List A, Gore SD, Seymour JF, Bennett JM, Byrd J, Backstrom J, Zimmerman L, McKenzie D, Beach C, Silverman LR; International Vidaza High-Risk MDS Survival Study Group. Efficacy of azacitidine compared with that of conventional care regimens in the treatment of higher-risk myelodysplastic syndromes: a randomised, open-label, phase III study. Lancet Oncol. 2009 Mar;10(3):223-32. doi: 10.1016/S1470-2045(09)70003-8. Epub 2009 Feb 21. PMID 19230772
- [Background] Fenaux P, Giagounidis A, Selleslag D, Beyne-Rauzy O, Mufti G, Mittelman M, Muus P, Te Boekhorst P, Sanz G, Del Canizo C, Guerci-Bresler A, Nilsson L, Platzbecker U, Lubbert M, Quesnel B, Cazzola M, Ganser A, Bowen D, Schlegelberger B, Aul C, Knight R, Francis J, Fu T, Hellstrom-Lindberg E; MDS-004 Lenalidomide del5q Study Group. A randomized phase 3 study of lenalidomide versus placebo in RBC transfusion-dependent patients with Low-/Intermediate-1-risk myelodysplastic syndromes with del5q. Blood. 2011 Oct 6;118(14):3765-76. doi: 10.1182/blood-2011-01-330126. Epub 2011 Jul 13. PMID 21753188
- [Background] Mallo M, Luno E, Sanzo C, Cervera J, Haase D, Schanz J, Garcia-Manero G, del Canizo C, Sanz GF, Sole F. Clinical impact of the clone size in MDS cases with monosomy 7 or 7q deletion, trisomy 8, 20q deletion and loss of Y chromosome. Leuk Res. 2011 Jun;35(6):834-6. doi: 10.1016/j.leukres.2011.01.003. Epub 2011 Jan 26. PMID 21269692
- [Background] Della Porta MG, Galli A, Bacigalupo A, Zibellini S, Bernardi M, Rizzo E, Allione B, van Lint MT, Pioltelli P, Marenco P, Bosi A, Voso MT, Sica S, Cuzzola M, Angelucci E, Rossi M, Ubezio M, Malovini A, Limongelli I, Ferretti VV, Spinelli O, Tresoldi C, Pozzi S, Luchetti S, Pezzetti L, Catricala S, Milanesi C, Riva A, Bruno B, Ciceri F, Bonifazi F, Bellazzi R, Papaemmanuil E, Santoro A, Alessandrino EP, Rambaldi A, Cazzola M. Clinical Effects of Driver Somatic Mutations on the Outcomes of Patients With Myelodysplastic Syndromes Treated With Allogeneic Hematopoietic Stem-Cell Transplantation. J Clin Oncol. 2016 Oct 20;34(30):3627-3637. doi: 10.1200/JCO.2016.67.3616. PMID 27601546
- [Background] Gerstung M, Pellagatti A, Malcovati L, Giagounidis A, Porta MG, Jadersten M, Dolatshad H, Verma A, Cross NC, Vyas P, Killick S, Hellstrom-Lindberg E, Cazzola M, Papaemmanuil E, Campbell PJ, Boultwood J. Combining gene mutation with gene expression data improves outcome prediction in myelodysplastic syndromes. Nat Commun. 2015 Jan 9;6:5901. doi: 10.1038/ncomms6901. PMID 25574665
- [Background] Gerstung M, Papaemmanuil E, Martincorena I, Bullinger L, Gaidzik VI, Paschka P, Heuser M, Thol F, Bolli N, Ganly P, Ganser A, McDermott U, Dohner K, Schlenk RF, Dohner H, Campbell PJ. Precision oncology for acute myeloid leukemia using a knowledge bank approach. Nat Genet. 2017 Mar;49(3):332-340. doi: 10.1038/ng.3756. Epub 2017 Jan 16. PMID 28092685
- [Background] Schneider RK, Adema V, Heckl D, Jaras M, Mallo M, Lord AM, Chu LP, McConkey ME, Kramann R, Mullally A, Bejar R, Sole F, Ebert BL. Role of casein kinase 1A1 in the biology and targeted therapy of del(5q) MDS. Cancer Cell. 2014 Oct 13;26(4):509-20. doi: 10.1016/j.ccr.2014.08.001. Epub 2014 Sep 18. PMID 25242043
- [Background] Platzbecker U, Germing U, Gotze KS, Kiewe P, Mayer K, Chromik J, Radsak M, Wolff T, Zhang X, Laadem A, Sherman ML, Attie KM, Giagounidis A. Luspatercept for the treatment of anaemia in patients with lower-risk myelodysplastic syndromes (PACE-MDS): a multicentre, open-label phase 2 dose-finding study with long-term extension study. Lancet Oncol. 2017 Oct;18(10):1338-1347. doi: 10.1016/S1470-2045(17)30615-0. Epub 2017 Sep 1. PMID 28870615
- [Background] Platzbecker U, Hofbauer LC, Ehninger G, Holig K. The clinical, quality of life, and economic consequences of chronic anemia and transfusion support in patients with myelodysplastic syndromes. Leuk Res. 2012 May;36(5):525-36. doi: 10.1016/j.leukres.2012.01.006. Epub 2012 Feb 1. PMID 22300879
- [Background] Platzbecker U, Schetelig J, Finke J, Trenschel R, Scott BL, Kobbe G, Schaefer-Eckart K, Bornhauser M, Itzykson R, Germing U, Beelen D, Ehninger G, Fenaux P, Deeg HJ, Ades L; German MDS Study; Cooperative Transplant Study Group; Fred Hutchinson Cancer Research Center; Groupe Francophone des Myelodysplasies. Allogeneic hematopoietic cell transplantation in patients age 60-70 years with de novo high-risk myelodysplastic syndrome or secondary acute myelogenous leukemia: comparison with patients lacking donors who received azacitidine. Biol Blood Marrow Transplant. 2012 Sep;18(9):1415-21. doi: 10.1016/j.bbmt.2012.05.003. Epub 2012 May 11. PMID 22579634
- [Background] Park S, Hamel JF, Toma A, Kelaidi C, Thepot S, Campelo MD, Santini V, Sekeres MA, Balleari E, Kaivers J, Sapena R, Gotze K, Muller-Thomas C, Beyne-Rauzy O, Stamatoullas A, Kotsianidis I, Komrokji R, Steensma DP, Fensterl J, Roboz GJ, Bernal T, Ramos F, Calabuig M, Guerci-Bresler A, Bordessoule D, Cony-Makhoul P, Cheze S, Wattel E, Rose C, Vey N, Gioia D, Ferrero D, Gaidano G, Cametti G, Pane F, Sanna A, Germing U, Sanz GF, Dreyfus F, Fenaux P. Outcome of Lower-Risk Patients With Myelodysplastic Syndromes Without 5q Deletion After Failure of Erythropoiesis-Stimulating Agents. J Clin Oncol. 2017 May 10;35(14):1591-1597. doi: 10.1200/JCO.2016.71.3271. Epub 2017 Mar 28. PMID 28350519
- [Background] Lamarque M, Raynaud S, Itzykson R, Thepot S, Quesnel B, Dreyfus F, Rauzy OB, Turlure P, Vey N, Recher C, Dartigeas C, Legros L, Delaunay J, Visanica S, Stamatoullas A, Fenaux P, Ades L. The revised IPSS is a powerful tool to evaluate the outcome of MDS patients treated with azacitidine: the GFM experience. Blood. 2012 Dec 13;120(25):5084-5. doi: 10.1182/blood-2012-09-453555. No abstract available. PMID 23243156
- [Background] Itzykson R, Thepot S, Quesnel B, Dreyfus F, Beyne-Rauzy O, Turlure P, Vey N, Recher C, Dartigeas C, Legros L, Delaunay J, Salanoubat C, Visanica S, Stamatoullas A, Isnard F, Marfaing-Koka A, de Botton S, Chelghoum Y, Taksin AL, Plantier I, Ame S, Boehrer S, Gardin C, Beach CL, Ades L, Fenaux P; Groupe Francophone des Myelodysplasies(GFM). Prognostic factors for response and overall survival in 282 patients with higher-risk myelodysplastic syndromes treated with azacitidine. Blood. 2011 Jan 13;117(2):403-11. doi: 10.1182/blood-2010-06-289280. Epub 2010 Oct 12. PMID 20940414
- [Background] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Gattermann N, Germing U, Sanz G, List AF, Gore S, Seymour JF, Dombret H, Backstrom J, Zimmerman L, McKenzie D, Beach CL, Silverman LR. Azacitidine prolongs overall survival compared with conventional care regimens in elderly patients with low bone marrow blast count acute myeloid leukemia. J Clin Oncol. 2010 Feb 1;28(4):562-9. doi: 10.1200/JCO.2009.23.8329. Epub 2009 Dec 21. PMID 20026804
- [Background] Mallo M, Del Rey M, Ibanez M, Calasanz MJ, Arenillas L, Larrayoz MJ, Pedro C, Jerez A, Maciejewski J, Costa D, Nomdedeu M, Diez-Campelo M, Lumbreras E, Gonzalez-Martinez T, Marugan I, Such E, Cervera J, Cigudosa JC, Alvarez S, Florensa L, Hernandez JM, Sole F. Response to lenalidomide in myelodysplastic syndromes with del(5q): influence of cytogenetics and mutations. Br J Haematol. 2013 Jul;162(1):74-86. doi: 10.1111/bjh.12354. Epub 2013 Apr 25. PMID 23614682
- [Background] Mekinian A, Grignano E, Braun T, Decaux O, Liozon E, Costedoat-Chalumeau N, Kahn JE, Hamidou M, Park S, Puechal X, Toussirot E, Falgarone G, Launay D, Morel N, Trouiller S, Mathian A, Gombert B, Schoindre Y, Lioger B, De Wazieres B, Amoura Z, Buchdaul AL, Georgin-Lavialle S, Dion J, Madaule S, Raffray L, Cathebras P, Piette JC, Rose C, Ziza JM, Lortholary O, Montestruc F, Omouri M, Denis G, Rossignol J, Nimubona S, Ades L, Gardin C, Fenaux P, Fain O. Systemic inflammatory and autoimmune manifestations associated with myelodysplastic syndromes and chronic myelomonocytic leukaemia: a French multicentre retrospective study. Rheumatology (Oxford). 2016 Feb;55(2):291-300. doi: 10.1093/rheumatology/kev294. Epub 2015 Sep 8. PMID 26350487
- [Background] Fraison JB, Mekinian A, Grignano E, Kahn JE, Arlet JB, Decaux O, Denis G, Buchdahl AL, Omouri M, Maigne G, Aouba A, Leon N, Berthier S, Liozon E, Park S, Gardin C, Lortholary O, Rossignol J, Fenaux P, Fain O, Braun T. Efficacy of Azacitidine in autoimmune and inflammatory disorders associated with myelodysplastic syndromes and chronic myelomonocytic leukemia. Leuk Res. 2016 Apr;43:13-7. doi: 10.1016/j.leukres.2016.02.005. Epub 2016 Feb 20. PMID 26922775
- [Background] Khaznadar Z, Boissel N, Agaugue S, Henry G, Cheok M, Vignon M, Geromin D, Cayuela JM, Castaigne S, Pautas C, Raffoux E, Lachuer J, Sigaux F, Preudhomme C, Dombret H, Dulphy N, Toubert A. Defective NK Cells in Acute Myeloid Leukemia Patients at Diagnosis Are Associated with Blast Transcriptional Signatures of Immune Evasion. J Immunol. 2015 Sep 15;195(6):2580-90. doi: 10.4049/jimmunol.1500262. Epub 2015 Aug 5. PMID 26246143